CLINICAL TRIAL: NCT04577365
Title: Validation of a New Scale of Balance Recovery Confidence for Community-dwelling Older Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Queen Margaret University (Other)
Collaborators: Singapore Institute of Technology (Other)
Responsible Party: Principal Investigator, Shawn Leng-Hsien Soh, Principal Investigator, Queen Margaret University
Other Study IDs: REP0220
Record Dates: First submitted 2020-09-30; First posted 2020-10-06 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Fall; Self Efficacy
Keywords: Accidental Falls; patient outcome assessment; postural balance; self-efficacy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction: Patient-reported outcome measures (PROMs) provide clinicians with a greater understanding of patients' perceived ability in their physical performance. Existing PROMs on falls efficacy provide meaningful information about the perceived ability in older people to perform common activities of daily living without falling. However, the perceived ability to recover the balance from a slip, a trip, or volitional movements has been inadequately assessed. Balance recovery confidence relates to the judgement of self-reactive ability. The scale of balance recovery confidence (BRC) is a new PROM that measures perceived balance recovery self-efficacy. The purpose of the study protocol is to describe the first psychometric evaluation of BRC's measurement properties.

Methods and analysis: This study is a validation phase of a newly developed PROM conducted in Singapore. Two hundred community-dwelling older adults, aged 65 years and older, will complete five self-reported instruments (BRC), Activities-specific Balance Confidence Scale (ABC), Falls Efficacy Scale-International (FES-I), Late-Life Function and Disability Instrument-Function (LLDI-F) and Global Perceived Effect (GPE) and three performance measures (Hand strength dynamometer, 30-second Chair Stand, Mini BESTest). Classical test theory methods will assess acceptability, data completeness, targeting of the items, scaling assumptions, internal consistency reliability and construct validity. Factor analysis will establish unidimensionality. Rasch analysis will evaluate item fit, differential item functioning, response scale ordering, targeting of persons and items and the reliability.

DETAILED DESCRIPTION:
Introduction: This study aims to conduct the first evaluation of measurement properties in the scale of balance recovery confidence. There are several measurement properties such as unidimensionality, validity (to what extent does the instrument measure the construct it purports to measure) and reliability (the degree to which measurement is free from error) of the PROM that is needed to be studied.

This psychometric validation aims to provide evidence that the PROM can be purposefully used in practice, given that rigorous methods have been applied for the development and validation of the BRC. For the study, balance recovery confidence is defined as the perceived ability to recover one's balance from perturbations, such as a slip, a trip, or a loss of balance that can occur in common, everyday activities. This focus will leave little ambiguity about precisely what is being measured. The resulting questionnaire is intended to be approximately 20 questions and should not take longer than 10 min to complete. The instrument is not intended to be used as a diagnostic tool of impaired specific balance recovery mechanisms. The BRC allows clinicians and researchers to quantifiably determine the balance recovery confidence in older adults and use the scale as a conduit for understanding older people's perspectives when encountering different perturbations during their daily activities.

The objectives are to:

1. To evaluate the measurement properties of the BRC, i.e. acceptability, targeting, scaling assumptions and reliability using Classical Test Theory (CTT), the internal scale structure using Rasch measurement theory in the Singapore community-dwelling older adults.
2. To assess the construct validity of the refined BRC against commonly used PROMs and performance measures in the Singapore community-dwelling older adults.
3. To refine the items, response categories, and scale structure of the BRC using Rasch measurement theory in an English-speaking sample of community-dwelling older adults in Singapore.

Methods: Participants will attend two sessions in the study. In the first session, the researcher will use a measurement data form to record the participants' results of four questionnaires: BRC, ABC, FES-I, LLFDI-F and three performance measures: Jamar hand strength dynamometer, 30-second chair stand test and Mini BESTest. After seven days, participants will attend the second session to complete the BRC, and the GPE scale which will be used to ensure participants' perception of their abilities remained unchanged during the seven days. The time interval of 7-day had been reported to be sufficient to minimise recall bias. Participants will be asked if they have had experienced a fall, near-fall, or encountered any incident that might affect their balance recovery ability over the past seven days.

Statistical analysis: Quantitative data will be analysed and interpreted through two measurement test theories using IBM SPSS Statistic V.26.0 and Winsteps V.4.5.0. Classical test theory is a traditional quantitative approach to test the validity and reliability of a scale based on its items. This approach is based on the assumption that every observed score is a function of an individual's true score and random error. In contrast, RA works on the probability of a person's level on an item is a function of the person's ability and of the difficulty of the item. RA evaluates a scale against a mathematical measurement model and analyses the scale at the level of each item, and each person. Measurement properties including unidimensionality, internal structure, validity and reliability will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 65-years and older,
* Living in the community,
* Functionally independent with or without the use of a walking aid and be able to read,
* Write and communicate in English.

Exclusion Criteria:

* Require any physical assistance from another person to walk within the home,
* Presenting with clinical observable severe cognitive impairment.
* Unable to provide written consent to participate in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Scale of Balance Recovery Confidence | 5 minutes
  The scale of balance recovery confidence measures the perceived balance recovery self-efficacy in community-dwelling older adults. A response option ranged from 0 to 10 is listed with 10 indicating "Highly certain can do" and 0 refers to "Cannot do at all". The outcome measure is administered on Day 1 and Day 7.
Activities-specific Balance Confidence Scale | 5 minutes
  The Activities-specific Balance Confidence scale assesses older adults' confidence that they will not fall or lose their balance when performing several progressively challenging balance and mobility tasks. The response option ranged from 0% (no confidence) to 100% (complete confidence). The outcome measure is administered on Day 1
Falls Efficacy Scale - International | 5 minutes
  The Falls Efficacy Scale- International measures fear of falling or "concerns about falling" relating to basic and more demanding activities both physical and social. The response option ranged from 1-4 depicted by 1 for being not at all concerned, 2 for being somewhat concerned, 3 for being fairly concerned and 4 for being very concerned. The outcome measure is administered on Day 1
Late-Life Function and Disability Instrument-Function component | 5 minutes
  The Late-Life Function and Disability Instrument-Functional component of the instrument evaluates self-reported difficulty a person has in performing activities of daily living tasks. Factors that may influence the difficulty in task performance include pain, fatigue, fear, weakness, soreness, ailment, health conditions, and disabilities.There are 32 items with response options of "none," "a little," "some," "quite a lot," and "cannot do." An additional eight items will be completed by those who use canes or walkers. The outcome measure is administered on Day 1

SECONDARY OUTCOMES:
Jamar hand strength dynamometer | 10 minutes
  The handheld dynamometer provides a quantitative measure of isometric grip strength of the hand by determining the amount of static force that the hand can squeeze around a dynamometer. The outcome measure is administered on Day 1
30-second chair stand test | 10 minutes
  A quantitative measure used as test functional lower extremity strength as well as to obtain an indicator of functional independence with repeated performance of sit to stand from a chair within 30 seconds. The outcome measure is administered on Day 1
Mini BESTest | 10 minutes
  The Mini BESTest assesses "anticipatory postural adjustment", "postural responses", "sensory orientation" and "balance during gait". The outcome measure is administered on Day 1.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Soh, Principal Investigator — Singapore Institute of Technology
Locations (1):
- Singapore Institute of Technology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be shared
Supporting Information: Study Protocol
Time Frame: The study protocol will be made available after publication
Access Criteria: - PROM developers

REFERENCES:
- [Background] Tokur D, Grimmer M, Seyfarth A. Review of balance recovery in response to external perturbations during daily activities. Hum Mov Sci. 2020 Feb;69:102546. doi: 10.1016/j.humov.2019.102546. Epub 2019 Dec 31. PMID 31989948
- [Background] Tinetti ME, Richman D, Powell L. Falls efficacy as a measure of fear of falling. J Gerontol. 1990 Nov;45(6):P239-43. doi: 10.1093/geronj/45.6.p239. PMID 2229948
- [Background] Powell LE, Myers AM. The Activities-specific Balance Confidence (ABC) Scale. J Gerontol A Biol Sci Med Sci. 1995 Jan;50A(1):M28-34. doi: 10.1093/gerona/50a.1.m28. PMID 7814786
- [Background] Simpson JM, Worsfold C, Fisher KD, Valentine JD. The CONFbal scale: a measure of balance confidence--a key outcome of rehabilitation. Physiotherapy. 2009 Jun;95(2):103-9. doi: 10.1016/j.physio.2008.12.004. Epub 2009 Mar 24. PMID 19627691
- [Background] Horak FB, Wrisley DM, Frank J. The Balance Evaluation Systems Test (BESTest) to differentiate balance deficits. Phys Ther. 2009 May;89(5):484-98. doi: 10.2522/ptj.20080071. Epub 2009 Mar 27. PMID 19329772
- [Background] Jette AM, Haley SM, Coster WJ, Kooyoomjian JT, Levenson S, Heeren T, Ashba J. Late life function and disability instrument: I. Development and evaluation of the disability component. J Gerontol A Biol Sci Med Sci. 2002 Apr;57(4):M209-16. doi: 10.1093/gerona/57.4.m209. PMID 11909885
- [Background] Kamper SJ, Ostelo RW, Knol DL, Maher CG, de Vet HC, Hancock MJ. Global Perceived Effect scales provided reliable assessments of health transition in people with musculoskeletal disorders, but ratings are strongly influenced by current status. J Clin Epidemiol. 2010 Jul;63(7):760-766.e1. doi: 10.1016/j.jclinepi.2009.09.009. Epub 2010 Jan 8. PMID 20056385